CLINICAL TRIAL: NCT00326066
Title: A Study of the Trabecular Micro-bypass Stent in Combination With Cataract Surgery in Subjects With Newly Diagnosed Open Angle Glaucoma and Subjects Diagnosed With Ocular Hypertension
Brief Title: A Study of the iStent in Combo With Cataract Surgery in Newly Diagnosed Open Angle Glaucoma or OH Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCF-007
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Open-Angle Glaucoma
Keywords: Open angle; Glaucoma; Surgery; Cataract
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Device: Glaucoma Surgery
- 2 (Placebo Comparator)
  Interventions: Procedure: cataract surgery only

INTERVENTIONS:
Device: Glaucoma Surgery — Comparing the effect in reducing IOP with two Trabecular Bypass Microstents Versus none in patients undergoing cataract surgery, with early open angle glaucoma or ocular hypertension.
  Other Names: two Glaukos iStent Trabecular Bypass Microstents
  Arms: 1
Procedure: cataract surgery only — Subjects will undergo routine cataract surgery only (no stent implant).
  Other Names: Phacoemulsification
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the iStent trabecular micro-bypass stent in reducing intraocular pressure (IOP) in subjects with newly diagnosed open-angle glaucoma and subjects diagnosed with Ocular hypertension.

DETAILED DESCRIPTION:
The study will compare the reduction in IOP of those subjects implanted with two Glaukos micro-stents with the reduction in IOP for patients receiving only primary medical therapy (Xalatan - Latanoprost) or cataract surgery alone. Both groups will undergo routine cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with open-angle glaucoma (OAG) or Ocular Hypertension with subjects not yet taking any glaucoma medications or recently diagnosed with mild open-angle glaucoma and are currently being treated with up to 2 glaucoma medications.
* All subjects must need cataract surgery.

Exclusion Criteria:

* Angle closure glaucoma
* Secondary glaucomas except pseudoexfoliative and pigmentary; no neovascular, uveitic or angle recession glaucoma
* Prior glaucoma procedures (eg trabeculectomy, viscocanalostomy, ALT, SLT, shunt implant, collagen implant, cyclo destructive procedures etc)
* Fellow eye already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Efficacy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Affairs, Study Director — Glaukos Corporation
Locations (9):
- Vienna Medical Hospital, Vienna, Austria
- Germany (3):
  - Mainz University, Mainz
  - Augenklinik der Technischen Universitat, Munich
  - Universitats- Augenklinik, Würzburg
- Netherlands (2):
  - The Netherlands Ophthalmic Research Institute, Amsterdam
  - Ophthalmic Clinic, Rotterdam
- Spain (2):
  - Clinico San Carlos, Madrid
  - Instituto Oftalmológico de Aragón, Zaragoza
- Beyoglu Eye Research and Education Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Fernandez-Barrientos Y, Garcia-Feijoo J, Martinez-de-la-Casa JM, Pablo LE, Fernandez-Perez C, Garcia Sanchez J. Fluorophotometric study of the effect of the glaukos trabecular microbypass stent on aqueous humor dynamics. Invest Ophthalmol Vis Sci. 2010 Jul;51(7):3327-32. doi: 10.1167/iovs.09-3972. Epub 2010 Mar 5. PMID 20207977